CLINICAL TRIAL: NCT02192983
Title: A Comparison of XELOX Regimen and EOX Regimen as Neoadjuvant Chemotherapy Regimen for Locally Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Tianshu Liu (Other)
Responsible Party: Sponsor-Investigator, Tianshu Liu, Chairman of the department of oncology, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: zswy002
Record Dates: First submitted 2014-07-15; First posted 2014-07-17 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Locally Advanced Gastric Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chemotherapy regimen: those with XELOX regimen and those with EOX regimen

SUMMARY:
This study is designed to assess what is the better neoadjuvant chemotherapy regimen for patients with initially unresectable locally advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* more than 2 regional bulky lymph nodes macroscopic tumor type is either the Borrmann type 4 or large type 3 tumor invades adjacent structures (T4b)

Exclusion Criteria:

* peritoneal metastasis confirmed by CT scan lung metastasis, liver metastasis, pleural effusion, and/or other distant metastasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 242
Sampling Method: Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2008-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: tianshu liu, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Ethics Committee, Shanghai, Shanghai Municipality, China